CLINICAL TRIAL: NCT03346200
Title: A Randomised, Double Blinded, Six-armed Placebo Controlled Study to Investigate Optimal Dose of Tamoxifen With the Most Favourable Side Effect Spectre and With Mammography Density Reduction Non-inferior to That of 20 mg Tamoxifen
Brief Title: Low Dose Tamoxifen for Mammographic Density Reduction
Acronym: KARISMA2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Per Hall (Other)
Responsible Party: Sponsor-Investigator, Per Hall, Professor, MD, PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016-000882-22
Record Dates: First submitted 2017-11-01; First posted 2017-11-17 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Risk Reduction; Mammographic Density Reduction
Keywords: Breast cancer; Prevention; Tamoxifen
MeSH Terms: conditions — Risk Reduction Behavior; Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- 20 mg tamoxifen (Active Comparator)
  Interventions: Drug: Tamoxifen Oral Tablet
- 10 mg tamoxifen (Experimental)
  Interventions: Drug: Tamoxifen Oral Tablet
- 5 mg tamoxifen (Experimental)
  Interventions: Drug: Tamoxifen Oral Tablet
- 2.5 mg tamoxifen (Experimental)
  Interventions: Drug: Tamoxifen Oral Tablet
- 1 mg tamoxifen (Experimental)
  Interventions: Drug: Tamoxifen Oral Tablet
- 0 mg tamoxifen (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Tamoxifen Oral Tablet — Randomised dose of tamoxifen 1 pill/day for 180 days
  Arms: 1 mg tamoxifen; 10 mg tamoxifen; 2.5 mg tamoxifen; 20 mg tamoxifen; 5 mg tamoxifen
Drug: Placebo Oral Tablet — Randomised dose of tamoxifen 1 pill/day for 180 days
  Arms: 0 mg tamoxifen

SUMMARY:
KARISMA2 is a randomized, double-blinded, six-armed placebo controlled study to identify a low dose of tamoxifen, with less side-effects and a density reduction non-inferior to the standard dose of 20 mg.

DETAILED DESCRIPTION:
This is a dose determination study aiming to identify the optimal tamoxifen dose for reducing the risk of breast cancer. The change in mammographic density is a very good marker of therapy response. Investigators will test if 1 mg, 2.5 mg, 5 mg and 10 mg reduce the mammographic density to the same extent as 20 mg.

1440 healthy women 40-74 yrs were included when adhering the national Swedish mammography screening program between 2016- 2019. Women were randomized and treated daily for 6 months. Mammograms were taken at baseline and at end of treatment and side effects were measured throughout the study trough schedueled questionnaires and spontaneous AE-reporting.

ELIGIBILITY:
Inclusion Criteria:

* Attending the national mammography screening program, i.e. aged 40-74 and has performed a screening mammogram maximum 3 months prior to study inclusion
* Having a measurable mammographic density, i.e. ≥4.5 % density (volumetric) measured by Volpara
* Informed consent must be signed before any study specific assessments have been performed

Exclusion Criteria:

* Pregnancy at start, during time of study medication and up to 3 months after quitting study medication
* Breast feeding at start, during time of study medication and up to 3 months after quitting study medication
* Any previous or current diagnosis of breast cancer (including carcinoma in situ)
* Mammographic BI-RADS code 3 or above at baseline mammography, or at a diagnostic mammography during time of treatment (the first 6 months of the study)
* Any previous diagnosis of cancer with the exception of non-melanoma skin cancer and in situ cancer of the cervix
* Currently using oral oestrogen and progesterone based hormone replacement therapy
* Current use of hormone contraceptive with hormones, e.g. hormonal contraceptive pills, or progesterone implants. Hormonal intrauterine devices are accepted.
* A history of thrombo-embolic disease such as embolies, deep vein thrombosis, stroke, TIA or cardiac arrest.
* Known APC (Activated protein C )- resistance, an inherited hemostatic disorder
* A history of major surgery of the breast, e.g. reduction or enlargement, which might affect density measurements
* Women who have an increased risk of venous thrombosis due to immobilization, e.g. using wheelchair
* Known uncontrolled diabetes
* Hypertension at baseline, defined as systolic pressure higher than 140 mm Hg and diastolic higher than 90 mm Hg
* Use of drugs that interfere with CYP2D6 expression such as Seroxat (paroxetine), Fontex (fluoxetin) and Zyban / Voxra (bupropion)
* Use of Waran (warfarin)
* Non-medical approved drugs against hot-flashes including phytooestrogen
* Not able to understand study information and/or informed consent

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female mammography screening population in Sweden age 40-74
Enrollment: 1440 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Hall, Professor, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eriksson M, Eklund M, Borgquist S, Hellgren R, Margolin S, Thoren L, Rosendahl A, Lang K, Tapia J, Backlund M, Discacciati A, Crippa A, Gabrielson M, Hammarstrom M, Wengstrom Y, Czene K, Hall P. Low-Dose Tamoxifen for Mammographic Density Reduction: A Randomized Controlled Trial. J Clin Oncol. 2021 Jun 10;39(17):1899-1908. doi: 10.1200/JCO.20.02598. Epub 2021 Mar 18. PMID 33734864
- [Derived] Goransson S, Hernandez-Varas P, Hammarstrom M, Hellgren R, Backlund M, Lang K, Rosendahl AH, Eriksson M, Borgquist S, Stromblad S, Czene K, Hall P, Gabrielson M. Low-dose tamoxifen treatment reduces collagen organisation indicative of tissue stiffness in the normal breast: results from the KARISMA randomised controlled trial. Breast Cancer Res. 2024 Nov 26;26(1):163. doi: 10.1186/s13058-024-01919-1. PMID 39593191
- [Derived] Hammarstrom M, Gabrielson M, Crippa A, Discacciati A, Eklund M, Lundholm C, Backlund M, Wengstrom Y, Borgquist S, Bergqvist J, Eriksson M, Tapia J, Czene K, Hall P. Side effects of low-dose tamoxifen: results from a six-armed randomised controlled trial in healthy women. Br J Cancer. 2023 Jul;129(1):61-71. doi: 10.1038/s41416-023-02293-z. Epub 2023 May 6. PMID 37149701
- [Derived] Gabrielson M, Hammarstrom M, Backlund M, Bergqvist J, Lang K, Rosendahl AH, Borgquist S, Hellgren R, Czene K, Hall P. Effects of tamoxifen on normal breast tissue histological composition: Results from a randomised six-arm placebo-controlled trial in healthy women. Int J Cancer. 2023 Jun 1;152(11):2362-2372. doi: 10.1002/ijc.34430. Epub 2023 Jan 22. PMID 36637153
- See also: KARMA -Karolinska Mammography Project for Risk Prediction of Breast Cancer — https://karmastudy.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20 mg Tamoxifen | 10 mg Tamoxifen | 5 mg Tamoxifen | 2.5 mg Tamoxifen | 1 mg Tamoxifen | 0 mg Tamoxifen
Started | 241 | 243 | 240 | 235 | 239 | 242
Completed | 171 | 167 | 157 | 159 | 174 | 183
Not Completed | 70 | 76 | 83 | 76 | 65 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 mg Tamoxifen | 10 mg Tamoxifen | 5 mg Tamoxifen | 2.5 mg Tamoxifen | 1 mg Tamoxifen | 0 mg Tamoxifen | Total
Number analyzed (Participants) | 241 | 243 | 240 | 235 | 239 | 242 | 1440
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 181 | 179 | 185 | 181 | 193 | 177 | 1096
  >=65 years | 60 | 64 | 55 | 54 | 46 | 65 | 344
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (9.5) | 55.8 (10.0) | 55.1 (9.7) | 54.9 (9.7) | 54.3 (9.4) | 60.0 (9.9) | 55.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Only females included in this Breast cancer study
  Participants
    Female | 241 | 243 | 240 | 235 | 239 | 242 | 1440
    Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mammograpic Density Change
Description: Change in mammography density. In particular, we will test for noninferiority in the proportion of women in the intervention arms (placebo, 1 mg, 2.5 mg, 5 mg, 10 mg) who have a density reduction as great as or greater (after 6 months) than the median density reduction in the 20 mg arm.
Time Frame: 6 months treatment
Measure: Mean (95% Confidence Interval); unit: Percentage of change
Groups:
- 20 mg Tamoxifen; 10 mg Tamoxifen; 5 mg Tamoxifen; 2.5 mg Tamoxifen; 0 mg Tamoxifen: Randomised dose of tamoxifen 1 pill/day for 180 days. Primary outcome: Change in mammography density in relation to 20 mg (non-inferiority)
- 1 mg Tamoxifen: Randomised dose of tamoxifen 1 pill/day for 180 days.Primary outcome: Change in mammography density in relation to 20 mg (non-inferiority)
Arm/Group | 20 mg Tamoxifen | 10 mg Tamoxifen | 5 mg Tamoxifen | 2.5 mg Tamoxifen | 1 mg Tamoxifen | 0 mg Tamoxifen
Number analyzed (Participants) | 203 | 210 | 201 | 200 | 205 | 211
Percentage of change | -9.6 [-14.8 to -4.5] | -6.8 [-11.8 to -1.7] | -1.0 [-6.2 to 4.1] | -6.9 [-12.1 to -1.8] | -1.0 [-6.1 to 4.1] | 0.1 [-4.9 to 5.1]
Statistical Analysis 1: Comparison: 20 mg Tamoxifen; Test type: Non-Inferiority — The non-inferiority margin was based on the proportion of responders and was set to 17%. That is, we defined non-inferiority to mean that the proportion of responders in the non-referent study arms is not less than one third of the responders in the 20 mg group (50% minus 33% = 17%); p < 0.01, one-sided Wald tests; P-values were corrected for multiple comparisons using the Holm-Bonferroni method. Non-inferiority p-values were declared if less than a=0.025; Median Difference (Final Values) = 52.5, 97.5% CI 2-sided [41.9 to 100]

2. Secondary Outcome: Level of Side Effects
Description: Assess the level of side effects in the intervention arms compared to the 20 mg arm.
  Symptoms are reported on a 5-graded Likert score scale in a 48-item symptom questionnaire at Baseline and at End of treatment ( End of treatment= full-filled the 6 month treatment or at time of discontinuation prior to 6 months). The outcome measure is based on the sum in Likert score of five symptoms ('hot flashes', 'cold sweats', 'night sweats', 'vaginal discharge' and 'muscle cramps') which were found to have a significant change from start to the end of treatment in both pre- and postmenopausal women when contrasting the effect of 20 mg tamoxifen compared to women on placebo. The maximum/minimum range of change per symtom is 4 steps increase or decrease. Accordingly, in the Top-5 symtoms the maximum/minimum range is +/- 20. Higher scores mean a worse outcome.
Time Frame: From baseline (7-1days before first tablet) up to 6 months or day of discontionuation (prior to 6 months)
Population: In all 1175 women, whereof 454 (39%) premenopausal and 721 (61%) postmenopausal, constitute the per protocol population which fulfilled teh 48-item Symptom questionnaire at Baseline and at End of treatment (6month or at time of Early termination)
Measure: Mean (95% Confidence Interval); unit: Likert score change in Top5 Symptoms
Arm/Group | 20 mg Tamoxifen | 10 mg Tamoxifen | 5 mg Tamoxifen | 2.5 mg Tamoxifen | 1 mg Tamoxifen | 0 mg Tamoxifen
Number analyzed (Participants) | 199 | 199 | 188 | 194 | 193 | 202
Likert score change in Top5 Symptoms | 2.71 [2.29 to 3.13] | 2.97 [2.50 to 3.45] | 2.52 [2.07 to 2.97] | 2.39 [1.94 to 2.85] | 1.65 [1.24 to 2.06] | 0.36 [0.32 to 0.68]

3. Secondary Outcome: Drop Out Level
Description: Assess the level of drop out in the intervention arms compared to the 20 mg arm
Time Frame: From initiation of treatment (first tablet) up to 6 months of planned treatment (last tablet)
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | 20 mg Tamoxifen | 10 mg Tamoxifen | 5 mg Tamoxifen | 2.5 mg Tamoxifen | 1 mg Tamoxifen | 0 mg Tamoxifen
Number analyzed (Participants) | 241 | 242 | 240 | 235 | 239 | 242
Participants | 65 | 69 | 79 | 71 | 58 | 53

ADVERSE EVENTS:
Time Frame: From baseline (start of treatment) to end of study (6 months or early termination)
Description: Adverse events where collected through an app, by phone or email. Participants where urged to report when events occurred.
Arm/Group | 20 mg Tamoxifen | 10 mg Tamoxifen | 5 mg Tamoxifen | 2.5 mg Tamoxifen | 1 mg Tamoxifen | 0 mg Tamoxifen
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/243 | 0/240 | 0/235 | 0/239 | 0/242
Serious Adverse Events (participants affected / at risk) | 2/241 | 1/243 | 2/240 | 1/235 | 1/239 | 4/242
Other Adverse Events (participants affected / at risk) | 74/241 | 70/243 | 63/240 | 65/235 | 39/239 | 40/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg Tamoxifen (N=241) | 10 mg Tamoxifen (N=243) | 5 mg Tamoxifen (N=240) | 2.5 mg Tamoxifen (N=235) | 1 mg Tamoxifen (N=239) | 0 mg Tamoxifen (N=242)
Suspected TIA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Brain tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suspected Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg Tamoxifen (N=241) | 10 mg Tamoxifen (N=243) | 5 mg Tamoxifen (N=240) | 2.5 mg Tamoxifen (N=235) | 1 mg Tamoxifen (N=239) | 0 mg Tamoxifen (N=242)
Hot flush (Endocrine disorders) | 24 (34) | 32 (38) | 26 (47) | 25 (32) | 20 (21) | 13 (21)
Night sweats (Endocrine disorders) | 19 (42) | 21 (24) | 24 (49) | 22 (33) | 10 (17) | 13 (24)
Vaginal discharge (Endocrine disorders) | 18 (23) | 24 (35) | 21 (23) | 16 (23) | 8 (10) | 6 (7)
AE Free text (Endocrine disorders) | 36 (46) | 21 (22) | 17 (22) | 27 (30) | 15 (22) | 20 (22) — Unique reports not possible to cathegorize

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT03346200/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03346200/SAP_001.pdf